CLINICAL TRIAL: NCT03468569
Title: Relationship of Functional Movement Analysis With Injury History and Athletic Parameters In Handball Athletes
Brief Title: Functional Movement Analysis of Handball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Emre Serdar Vayvay, Lecturer, Medipol University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10840098-604.01.01-E.13036
Record Dates: First submitted 2017-11-01; First posted 2018-03-16 (Actual); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Injuries; Sports Physical Therapy
Keywords: Athletic Performance; Functional Movement Screen; Handball Athletes; Injury Prevention; Injury History
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Functional Movement Screen (Experimental): Movement Analysis for injury risk
  Interventions: Other: Functional Movement Screen
- Vertical Jump Test (Experimental): Jump test Height Measurement, Functional Movement Screen
  Interventions: Other: Functional Movement Screen
- Y Balance Test (Experimental): Functional lower extremity reach with balance, Functional Movement Screen
  Interventions: Other: Functional Movement Screen
- Illinois Agility Test (Experimental): Agility measurement, Functional Movement Screen
  Interventions: Other: Functional Movement Screen
- Injury History (No Intervention): Athletes injury history for last year was recorded as injury count.

INTERVENTIONS:
Other: Functional Movement Screen
  Arms: Functional Movement Screen; Illinois Agility Test; Vertical Jump Test; Y Balance Test

SUMMARY:
RELATIONSHIP OF FUNCTIONAL MOVEMENT ANALYSIS WITH INJURY HISTORY AND ATHLETIC PARAMETERS IN HANDBALL ATHLETES

Abstract Objectives: Handball is a popular sport in many countries. There is lack of knowledge about handball athlete's functional movement capacity. The aim of this study is to investigate the Functional Movement Screen (FMS™) scores, to evaluate the injury risks of handball athletes and to determine its relationship with athletic performance.

Design: Observational study. Methods: A total of 51 professional handball players in Turkey were included in this study. The sport-specific features and demographic data were recorded. The functional movement analysis was performed and agility and balance and force were evaluated.

DETAILED DESCRIPTION:
In august 2018, same evaluations will be done for same individuals.

ELIGIBILITY:
Inclusion Criteria:

* Become a team licensed handball athlete between ages 16-35
* Have not had a surgical operation involving the musculoskeletal system in the last six months
* Not having an obstacle to the realization of the tests to be carried out in the study
* Volunteering to participate in the work

Exclusion Criteria:

* If feeling any discomfort during the tests
* Do not want to go on study

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 51 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-05-18 (Actual); Study Completion 2017-05-18 (Actual)

PRIMARY OUTCOMES:
Functional Movement Screen Assessment (FMS) | 20 minutes
  0-21 (It has 7 subtests, and minimum 0 and maximum 3 is given for scoring.) Higher scores are better. For bilateral subtests, scoring is performed for both sides, and scoring is given according to lower side. ( Example; Right 2, Left 1 so 1 point score is given for that parameter. At last, all 7 scores summed for total score(0/21).

SECONDARY OUTCOMES:
Vertical Jump Test | 5 minutes
  Inches, Higher scores are better.
Y Balance Test | 10 minutes
  Functional Reach Measurement, higher scores are better.
Illinois Agility Test | 2 minutes
  Agility Measurement, Lower scores are better.

CONTACTS AND LOCATIONS:
Overall Officials: Devrim Tarakcı, PhD, Principal Investigator — Medipol University; Emre Serdar Vayvay, PhD, Study Director — Medipol University; Candan Algun, PhD,Prof, Study Chair — Medipol University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cook G, Burton L, Hoogenboom B. Pre-participation screening: the use of fundamental movements as an assessment of function - part 1. N Am J Sports Phys Ther. 2006 May;1(2):62-72. PMID 21522216
- [Background] Cook G, Burton L, Hoogenboom B. Pre-participation screening: the use of fundamental movements as an assessment of function - part 2. N Am J Sports Phys Ther. 2006 Aug;1(3):132-9. PMID 21522225
- [Background] Plisky PJ, Gorman PP, Butler RJ, Kiesel KB, Underwood FB, Elkins B. The reliability of an instrumented device for measuring components of the star excursion balance test. N Am J Sports Phys Ther. 2009 May;4(2):92-9. PMID 21509114
- [Background] Hachana Y, Chaabene H, Nabli MA, Attia A, Moualhi J, Farhat N, Elloumi M. Test-retest reliability, criterion-related validity, and minimal detectable change of the Illinois agility test in male team sport athletes. J Strength Cond Res. 2013 Oct;27(10):2752-9. doi: 10.1519/JSC.0b013e3182890ac3. PMID 23439329
- [Background] Raya MA, Gailey RS, Gaunaurd IA, Jayne DM, Campbell SM, Gagne E, Manrique PG, Muller DG, Tucker C. Comparison of three agility tests with male servicemembers: Edgren Side Step Test, T-Test, and Illinois Agility Test. J Rehabil Res Dev. 2013;50(7):951-60. doi: 10.1682/JRRD.2012.05.0096. PMID 24301432
- [Background] Carlock JM, Smith SL, Hartman MJ, Morris RT, Ciroslan DA, Pierce KC, Newton RU, Harman EA, Sands WA, Stone MH. The relationship between vertical jump power estimates and weightlifting ability: a field-test approach. J Strength Cond Res. 2004 Aug;18(3):534-9. doi: 10.1519/R-13213.1. PMID 15320676
- [Derived] Atalay ES, Tarakci D, Algun C. Are the functional movement analysis scores of handball players related to athletic parameters? J Exerc Rehabil. 2018 Dec 27;14(6):954-959. doi: 10.12965/jer.1836372.186. eCollection 2018 Dec. PMID 30656154